CLINICAL TRIAL: NCT01496859
Title: Observational Study of Baska Mask, a New Supraglottic Airway Device
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University College Hospital Galway (Other)
Responsible Party: Principal Investigator, John Laffey, Professor of Anaesthesia and Critical Care, Consultant Anaesthetist, University College Hospital Galway
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C.A.621
Record Dates: First submitted 2011-12-18; First posted 2011-12-21 (Estimated); Last update posted 2012-03-26 (Estimated); Status verified 2012-03

CONDITIONS: Performance and Safety of a New Supraglottic Airway Device
Keywords: Baska mask; supraglottic airway; airway management
MeSH Terms: interventions — Mutagenesis, Insertional

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Baska (Experimental)
  Interventions: Device: Placement and use of Baska mask

INTERVENTIONS:
Device: Placement and use of Baska mask — use of a supraglottic airway device as a standard part of a general anaesthetic
  Other Names: Baska mask

SUMMARY:
The Baska mask is a new supraglottic airway device . The investigators would like to assess its performance in setting in which the current standard - LMA device - is being used.

DETAILED DESCRIPTION:
Our group has performed a number of studies on novel airway devices. In this study we would like to evaluate a new supraglottic airway named Baska mask. We would like to monitor certain parameters (time to and ease of insertion, failure rate, seal pressures, complications etc) as regarding the performance and safety profile of this device. This is a descriptive case series of patients undergoing airway management under general anaesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Written informed Consent
* No relevant drug allergies
* Body-mass index (BMI) 20-35
* Age 18-65
* Non-urgent surgery of planned duration 0-2 hrs

Exclusion Criteria:

* Inability of patient/parent to understand or consent for the trial
* Non-English speakers
* Neck pathology
* Previous or anticipated problems with the upper airway or upper GI tract (reflux, hiatus hernia, oropharyngeal tumour, upper respiratory tract infection in the last 10 days etc)
* BMI >35
* Expected Difficult airway
* Live Pregnancy
* Increased risk for Gastric Aspiration

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-08; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Device Placement Success rate | within 30 mins of anaesthesia commencement
time to placement of device | within 30 mins of anaesthesia commencement
  from the moment the device touched until successful ventilation achieved or device removed

SECONDARY OUTCOMES:
airway leak pressure of the device | within 30 mins of anaesthetic commencement
user-rated ease of insertion of device | within 30 mins of anaestesia commencement
  10cm visual analog score to be used
complication rates | From the moment general anaesthesia commenced up to 1 day postoperatively
  complications specifically monitored will be desaturation episodes, laryngospasm, blood staining of the device, lip damage. We will record other complications related to the use of the device, including but not limited to loss of airway with need to manioulate mask/switch to alternative device, regurgitation, aspiration, teeth damage.
patient comfort indices | from the moment the patient awake up to 1 day postoperatively
  Throat pain, dysphagia and dysphonia will be assessed. 10 point verbal rating scale will be used

CONTACTS AND LOCATIONS:
Overall Officials: John G Laffey, FFARCSI, Principal Investigator — National University of Ireland, Galway and Galway University Hospitals
Locations (1):
- Galway University Hospitals, Galway, Galway, Ireland